CLINICAL TRIAL: NCT04527809
Title: Effect of Transcranial Direct Current Stimulation (tDCS) on a Virtual Reality Task in Individuals With Parkinson's Disease - Cross-sectional Project
Brief Title: Transcranial Direct Current Stimulation (tDCS) and Virtual Reality Task in Parkinson Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Talita Dias da Silva, Researcher, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02908218.0.0000.5390
Record Dates: First submitted 2020-08-02; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: The participants will undertake a single session of non-immersive VR tasks and tDCS-active or tDCS-sham.
Who Masked: Participant, Investigator
Masking Description: The participants, researchers and outcome assessors will remain blind throughout the study. To ensure proper blinding, the researcher responsible for that, will configurate the code of the tDCS device to sham or active before the proper application. It will be no difference between the devices for sham or active application of the tDCS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS-active (Experimental): tDCS-active will be performed over one session during the practice of VR games. The frequency of current applied will be 2mA. The stimulation intensity will be set at 100%, and the anodal electrode will be at the M1 area, and the cathodal electrode at the contralateral supraorbital area.
  Interventions: Device: tDCS-active
- tDCS-sham (Sham Comparator): tDCS-sham will be performed over one session during the practice of VR games. The frequency of current applied will be 2mA. The stimulation intensity will be set at 100%, and the anodal electrode will be at the M1 area, and the cathodal electrode at the contralateral supraorbital area. For the TDCS-sham the same active procedure setting will be used, however, the current will be interrupted after 20 seconds. This configuration will ensure that the electrical stimulus is interrupted before generating considerable stimuli, while the other characteristics of the intervention will be maintained.
  Interventions: Device: tDCS-sham

INTERVENTIONS:
Device: tDCS-active — One session of active Trasncranial Direct Current Stimulation combine to a Virtual Reality task.
  Arms: tDCS-active
Device: tDCS-sham — One session of sham Trasncranial Direct Current Stimulation combine to a Virtual Reality task.
  Arms: tDCS-sham

SUMMARY:
A double-blinded randomized controlled trial will be conducted, and all the participants will undertake one session of non-immersive VR tasks and tDCS-active or tDCS-sham. It will be a cross-sectional protocol. All protocol will have the assessment of Autonomic Nervous System, through Heart Rate Variability Analysis.

DETAILED DESCRIPTION:
Study Design: A double-blinded randomized controlled trial will be conducted, and all the participants will undertake a non-immersive VR tasks and tDCS-active or tDCS-sham. It will be a cross-sectional protocol.

Participants and sampling: Participants will be recruited through referral by the coordinators of places or institutions who has patients available to participate in the state of São Paulo-Brazil.

Inclusion Criteria: Participants with idiopathic Parkinson's Disease, with diagnosis previously confirmed by a specialized doctor, will be included if they have the agreement to participate in the research by signing the informed consent form.

Exclusion Criteria: Participants will be excluded if they used a wheelchair, were unable to complete the procedures due to any reported fatigue or due to having to leave previously, and who could not stand without any kind of help, such as a carrier or walking aids.

Randomization Participants: Participants will be randomly allocated to either group 1 (tDCS-active and VR tasks) or group 2 (tDCS-sham and VR tasks). Randomization will be under the control of a blinded investigator who will be the only person allowed to manage the electronic security file of the randomization to assign the individuals. The investigator will be blind to the group in which the participant is allocated to.

Blinding: The participants, researchers and outcome assessors will remain blind throughout the study. To ensure proper blinding, the researcher responsible for that, will configurate the code of the tDCS device to sham or active before the proper application. It will be no difference between the devices for sham or active application of the tDCS, because the same device has these two options.

Allocation concealment: Allocation concealment will successfully be reached since no one involved in this study (i.e. the participants, researchers, and outcome assessors) will be aware of the treatment allocations.

Intervention

All participants will attend the assigned tDCS and VR intervention as follows: there will be one session of application of tDCS and non-immersive VR tasks during twenty minutes of intervention. The researchers will be trained to perform all interventions tDCS-sham, tDCS-active and VR tasks.

Virtual Reality intervention

During the application of the tDCS-active or sham, it will be performed tasks in non-immersive virtual reality environment to stimulate and verify the performance in the timing coincident task present in the software that will be used provided by the "Bridge Games". A software developed by the Research and Technological Applications in Rehabilitation (Grupo de Pesquisa e Aplicação Tecnológica em Reabilitação - PATER) group of the School of Arts, Sciences, and Humanities of the University of Sao Paulo (EACH-USP).

Heart Rate Variability (HRV): It will be analyzed the HRV when the participant is already in the tDCS-active or sham application + VR task. The HRV analysis will follow the guidelines of the Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology (TFESC & NASPE, 1996). The strap (for data collection) will be positioned on the participant's chest, and the Polar RS800cx heart rate receiver will be positioned next to it. HRV will be recorded after the initial assessments at rest for 5 minutes, during virtual reality combined to tDCS training for 10 minutes and for rest after the intervention for 5 minutes, totalizing 20 minutes. For analysis of HRV data at rest 1000 consecutive RR intervals will be used and during the tasks 256 consecutive RR intervals will be used.

HR will be recorded beat by beat throughout the protocol by the Polar RS800CX FC Portable Monitor (Polar Electro, Finland) and RR intervals recorded by the monitor will be transferred to the Polar ProTreiner program (3.0 v., Polar Electro, Finland) , which allows HR visualization and cardiac period extraction in the "txt" file format.

Moderate digital filtering will be performed in the program itself complemented with manual filtering performed in Excel software to eliminate premature ectopic beats and artifacts, and only series with more than 95% sinus beats will be included in the study (Vanderlei et al., 2008).

HRV analysis will be performed using linear (time and frequency domain) and nonlinear methods that will be analyzed using Kubios HRV® software (Kubios HRV v.1.1 for Windows, Biomedical Signal Analysis Group, Department of Applied Physics, University of Kuopio, Finland).

tDCS Intervention

tDCS-active or tDCS-sham will be performed over one session during the practice of VR games. The frequency of current applied will be 2mA. The stimulation intensity will be set at 100%, and the anodal electrode will be at the M1 area, and the cathodal electrode at the contralateral supraorbital area. The device used will be the DS-Stimulator, from NeuroConn, which allows blindness of the subjects of the research and the experimenters.

Procedure: First, the demarcation and positioning of the tDCS device will be done, and the electrodes positioned at predetermined locations. Anodic TDCS with electrodes between 25-35 cm2, intensity of 2mA, density of up to 0.057 mA / cm2 for a period of 20 minutes will be used. However, for the TDCS-sham (placebo) the same active procedure setting will be used, however, the current will be interrupted after 20 seconds. This configuration will ensure that the electrical stimulus is interrupted before generating considerable stimuli, while the other characteristics of the intervention will be maintained.

After five minutes of stimulation at rest, the individuals performed the VR training with the MoveHero game, first with the upper limbs (during 5 minutes), then with the lower limbs (5 minutes). The participants will have the rest of the time (5 minutes) (with tDCS (sham or active). After each session the participant will be questioned about the presence of adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's Disease with diagnosis previoulsy confirmed by a specialized doctor.
* Agreement to participate in the research by signing the informed consent form.

Exclusion Criteria

* Wheelchair use
* Unable to complete the procedures due to any reported fatigue.
* Unable to complete the procedures due having to leave previously.
* Could not stand without any kind of help, such as a carrier or walking aids.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Motor skills improvement | 8 weeks.
  The motor skills will be analyzed through the games developed specifically for analysis of motor skills, such as (interception skills, speed, accuracy and reaction time).

SECONDARY OUTCOMES:
Heart Rate Variability | 8 weeks.
  The HRV will be analyzed at rest (20 minutes), during active/sham-tDCS (20 minutes) and during recover from the intervention (10 minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Talita D Silva, Ph.D., Principal Investigator — University of Sao Paulo
Locations (1):
- School of Arts, Sciences and Humanities of the University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No